CLINICAL TRIAL: NCT05377983
Title: The Effect of Lavender Oil Inhalation on Pain, Anxiety and Sleep Quality After Coronary Artery Bypass Graft: a Randomized Controlled Trial Protocol
Brief Title: The Effect of Lavender Oil Inhalation on Pain, Anxiety and Sleep Quality After Coronary Artery Bypass Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU-YDIKMEN-001
Record Dates: First submitted 2022-04-18; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: lavender oil; pain; anxiety; sleep
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Lavender oil inhalation will be performed by placing two drops of 2% lavender oil on a 5x5 cm sterile gauze cloth and asking the patient to smell it for three to five minutes.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): Lavender oil inhalation will be performed by placing two drops of 2% lavender oil on a 5x5 cm sterile gauze cloth and asking the patient to smell it for three to five minutes. Pain intensity and vital signs will be evaluated and recorded before each application and in the first five minutes after the application.
  Interventions: Other: Lavender oil inhalation will be performed by placing two drops of 2% lavender oil on a 5x5 cm sterile gauze cloth and asking the patient to smell it for three to five minutes
- the control group (No Intervention): The control group will only receive routine care.

INTERVENTIONS:
Other: Lavender oil inhalation will be performed by placing two drops of 2% lavender oil on a 5x5 cm sterile gauze cloth and asking the patient to smell it for three to five minutes — During the hospitalization period after CABG surgery, 2% lavender oil (Lavandula angustifolia) inhalation will be applied to the intervention group three times a day.
  Arms: the intervention group

SUMMARY:
Cardiovascular diseases are among the important health problems due to their increasing frequency and extensity in developed and developing countries. The most common method of treating cardiovascular diseases is Coronary Artery Bypass Graft (CABG) surgery. Common pain, sleep problems, and anxiety after CABG surgery can cause delay in postoperative recovery both physically and mentally. The study was planned to evaluate the effect of lavender oil inhalation on pain, anxiety level and sleep quality after CABG surgery.

DETAILED DESCRIPTION:
The study is a non-drug clinical, randomized controlled study, and will be conducted in the Cardiovascular Surgery Clinic of Bakırköy Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi associated to Istanbul Provincial Directorate of Health between December 2020 and December 2021. Criteria to be included in the study were determined as patients who are aged 18 years and over, underwent planned (elective) CABG surgery, whose lavender oil allergy test is negative, who is conscious with place, person and time orientation, who do not have any disability that would make communication difficult, can be communicated in Turkish, were informed to participate in the study and gave written consent. Criteria to be excluded from the study were determined as patients who are allergic to lavender, cosmetics and perfume, have a history of dermatitis, are diagnosed with sleep disorders and use any pharmacological and herbal medicines for these disorders, have sinusitis, upper respiratory tract infection, liver and kidney dysfunction, asthma and Chronic Obstructive Pulmonary Disease (COPD), whose blood pressure is not regulated, have arrhythmia, use controlled analgesia after surgery and cannot be communicated in Turkish. Criteria to be eliminated from the study were determined as patients, who have positive lavender oil allergy test, develop lavender allergy during application, want to leave the study voluntarily, and do not comply with the working process and conditions.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study were determined as follows:

  * 18 years of age or older,
  * undergoing elective CABG surgery,
  * negative lavender oil allergy test,
  * being conscious and oriented to place, person, and time,
  * not having any disability that would make communication difficult,
  * being able to communicate in Turkish, and
  * giving informed written consent to participate in the study.

Exclusion Criteria:

* The exclusion criteria for the study were determined as follows:

  * diagnosed with a sleep disorder or using any pharmacological and/or herbal medicine for insomnia,
  * being allergic to lavender, cosmetics, or perfume,
  * having a history of dermatitis,
  * sinusitis,
  * upper respiratory tract infection,
  * liver and kidney dysfunction,
  * asthma, and
  * chronic obstructive pulmonary disease,
  * not having regulated blood pressure,
  * having arrhythmia,
  * using patient-controlled analgesia after surgery,
  * not being able to communicate in Turkish.
* The remaining exclusion criteria were determined as follows:

  * a positive lavender oil allergy test,
  * development of lavender allergy during the study,
  * voluntarily deciding to leave the study, and
  * not complying with the study process and conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-08-24 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Up to five days
  Pain intensity, will be evaluated by NRS 3 times a day in the intervention and control group upon admission from the intensive care unit to the clinic, before and 30 minutes and four hours after each analgesic administration.In addition to this application, pain intensity will be evaluated with NRS before and five minutes after lavender oil inhalation in intervention group patients.
Anxiety level | Up to five days
  Anxitey level will be evaluated using the STAI-I at four hours after analgesic administration in the intervention group and at five minutes after lavender oil inhalation.
Sleep quality | Up to five days
  Sleep quality will also be evaluated using RCSQ every morning during.

CONTACTS AND LOCATIONS:
Overall Officials: YEŞİM DİKMEN AYDIN, Principal Investigator — Marmara University Faculty of Health Sciences,
Locations (1):
- Yesim Dikmen Aydin, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No